CLINICAL TRIAL: NCT05572983
Title: Phase Ⅱ Study of Chidamide in Combination With CHOP in Previously Untreated Peripheral T-Cell Lymphoma With Follicular Helper of T Cell Phenotype （SWIFT）
Brief Title: Phase Ⅱ Study of Chidamide in Combination With CHOP in Previously Untreated Peripheral T-Cell Lymphoma With Follicular Helper of T Cell Phenotype
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2022-485-02
Record Dates: First submitted 2022-09-30; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Peripheral T-Cell Lymphoma With Follicular Helper of T Cell Phenotype
MeSH Terms: interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Opiate Substitution Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide in Combination With CHOP (Experimental): Patients with previously untreated peripheral T-cell lymphoma with follicular helper of T cell phenotype will receive chidamide in combination with CHOP for 6 cycles (planned) (21 days per cycle). After 6 cycles of induction therapy, if complete remission (CR) was achieved, maintenance treatment with chidamide will be continued for two years.
  Interventions: Drug: Chidamide combined with CHOP; Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide combined with CHOP — A)Chidamide: 20mg, D1, 4,8,11, po; B) Cyclophosphamide: 750 mg/ m2, D1, iv.drip; C) Doxorubicin: 50 mg/ m2, D1, iv.drip (or epirubicin 70 mg/ m2, D1, iv.drip); D) Vincristine: 1.4 mg/ m2, D1 (maximum dose 2mg, maximum dose 1.5mg for age over 70 years), iv; E) Prednisone: 40mg/m2, D1-5,po
  Other Names: Induction treatment
Drug: Chidamide — Chidamide: 20mg，qw（d1,d4）,po
  Other Names: Maintenance treatment

SUMMARY:
This is a prospective, open-label, single arm, multicenter clinical study to evaluate the safety, tolerability, efficacy of chidamide in combination with CHOP in previously untreated peripheral T-cell lymphoma with follicular helper of T cell phenotype

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years old, male and female;
2. Peripheral T-Cell lymphoma with follicular helper of T cell phenotype confirmed by histopathology at the study center, including: ① Angioimmunoblastic T-cell lymphoma (AITL), ②follicular T-cell lymphoma (FTCL), and ③ other nodal PTCL with TFH phenotype;
3. Never received chemotherapy, radiotherapy, immunological and biological therapy for lymphoma before;
4. Autologous stem cell transplantation is not suitable or the patient refused to accept autologous stem cell transplantation;
5. There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma: measurable lesion: Positron emission tomography / computed tomography (PET/CT) or CT and/or MRI, intranode lesions with long diameter >1.5cm, short diameter >1.0cm, or exnode lesions with long diameter > 1.0 cm; PET CT examination of the lesion showing increased uptake in lymph nodes or extranodal areas (higher than liver) and imaging features consistent with lymphoma can be evaluated.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2；
7. Expected survival ≥ 3 months;
8. The following required baseline laboratory data:

   1. .White blood cell，WBC≥3.0×109/L(Bone marrow invasive patient≥2.0×109/L), Absolute neutrophil count，ANC ≥1.5×109/L, （Bone marrow invasive patient≥1.0×109/L), Platelet count (PLT) ≥75×109/L, （Bone marrow invasive patient≥50×109/L) ，Hemoglobin (HB)≥ 80g/L;
   2. .Total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN) (The liver invasion ≤3.0×ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN（The liver invasion≤5.0×ULN）
   3. .Renal function：creatinine, Cr≤1.5×ULN
   4. .Coagulation function： International Normalized Ratio (INR)≤1.5 ×ULN； Prothrombin Time (PT)、Activated Partial Thromboplastin Time (APTT)≤1.5×ULN（Unless the patient is receiving anticoagulant therapy and PT and APTT are within the expected range at screening time）；
   5. .Thyroid stimulating hormone (TSH) or free thyroid hormone (FT4) or free triiodothyronine (FT3) were within 10% of normal value (note: abnormal TSH caused by non-autoimmune causes can be included in the group);
9. Subjects fully understand and voluntarily participate in this study and sign informed consent

Exclusion Criteria:

1. A history of other malignant tumors within the past 5 years; Or other tumors (except basal cell carcinoma of the skin)
2. Patients with significant vital organ dysfunction;
3. Patients with active bleeding or newly developed thrombotic disease, and patients who are taking anticoagulants and having a bleeding tendency;
4. Patients with a known history of Human Immunodeficiency Virus (HIV) infection and/or acquired Immunodeficiency syndrome;
5. Patients with active chronic hepatitis B or active hepatitis C. Patients who are hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) or hepatitis C virus (HCV) antibody positive during the screening period require further testing for Hepatitis B Virus (HBV) DNA and HCV RNA. If HBV DNA is no more than 2500 copies /mL or 500 IU/mL and HCV RNA is no more than the lower limit of the assay, enrollment will be allowed after exclusion of treatment-requiring active hepatitis B or C infection. Hepatitis B virus carriers, stable hepatitis B (no more than 2500 copies /mL or 500 IU/mL of DNA) and cured hepatitis C patients were eligible;
6. Subjects who were treated with systemic glucocorticoids or other immunosuppressive agents for a condition within 14 days prior to initiation of study treatment {Local, ocular, intra-articular, intranasal, and inhaled glucocorticoids were allowed (with very low systemic absorption); Short-term (≤ 7 days) use of glucocorticoids for prophylactic treatment (e.g., contrast media allergy) or for treatment of non-autoimmune conditions (e.g., delayed hypersensitivity due to contact allergens) is allowed;
7. With active, and in the past two years need systemic treatment of autoimmune diseases (hormone replacement therapy is not considered a systemic treatment, such as type 1 diabetes, hypothyroidism only requiring thyroid hormone replacement therapy, low adrenocortical or pituitary function only requiring physiological doses of sugar cortical hormone replacement therapy ); Patients with autoimmune diseases that have not required systemic treatment in the past two years are eligible;
8. Patients with unstable angina and/or congestive heart failure or vascular disease (such as, the aortic aneurysm or peripheral venous thrombosis requiring surgery to repair) requiring hospital treatment within 12 months. Patients with other cardiac damage (such as poor control of arrhythmia, myocardial infarction, or ischemic) which may affect the drug safety evaluation within 12 months;
9. Patients who underwent major surgery within 28 days before enrollment; Less than 6 weeks after major organ surgery;
10. Long-term unhealed wounds or incomplete healing fractures;
11. Receive live attenuated vaccine (except influenza vaccine) within 4 weeks before enrollment or during the study period;
12. Pregnant or lactating women and subjects of reproductive age who do not want to take contraceptive measures;
13. Patients with mental illness or who cannot obtain informed consent;
14. There is active infection, except for tumor-related B symptoms and fever;
15. Cardiac clinical symptoms or diseases that are not well controlled, such as: I. Nyha grade 2 or above heart failure; II. Unstable angina pectoris; III. Myocardial infarction has occurred within 1 year; IV. Patients with clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
16. Ineligibility to participate in the study was determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | Up to 18 weeks
  Complete remission rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Objective response rate | Up to 18 weeks
  Objective Response rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
Partial remission rate | Up to 18 weeks
  Partial remission rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival（PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary antitumor efficacy
Overall survival | From date of randomization until the date of death from any cause, assessed up to 24 months
  To investigate the preliminary antitumor efficacy
Recurrence free survival | From date of randomization until the date ofthe occurrence of relapse or last visit, assessed up to 24 months
  To investigate the preliminary antitumor efficacy
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Up to 18 weeks
  To identify the incidence of AE and SAE

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University, Guangzhou, Guangdong, China